CLINICAL TRIAL: NCT01909609
Title: Parents' Knowledge and Perception of Benefits and Risks Regarding Neonatal Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Adam Eickmeyer, Senior Researcher, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HUM00073478
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Circumcision
Keywords: male

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Parent Survival Guide (Sham Comparator): This arm of the study will focus on the document that is normally given to all parents of newborn infants. It contains information on newborn care such as feeding, cleaning of the baby's penis, etc.
  Interventions: Other: Parent Survival Guide
- AAP Documents + Parent Survival Guide. (Experimental): This arm of the study will focus on documents created based off of the American Academy of Pediatrics 2012 policy statement. They contain information on the potential risks and benefits of neonatal circumcision. The Parent Survival Guide contains information on newborn care such as feeding, cleaning of the baby's penis, etc.
  Interventions: Other: AAP Documents; Other: Parent Survival Guide

INTERVENTIONS:
Other: AAP Documents
  Arms: AAP Documents + Parent Survival Guide.
Other: Parent Survival Guide

SUMMARY:
The American Academy of Pediatrics changed their stance on circumcision to "health benefits of newborn male circumcision outweigh the risks and that the procedure's benefits justify access to this procedure for families who choose it" (AAP, 2012).

We wonder if parents are aware of guidelines such as those of the AAP. Are parents able to make this medical decision by weighing the risks against the benefits of circumcision, or do they simply use sociocultural/religious reasons to make this decision? We hypothesize that parents are unaware of the specific benefits and risks of circumcision, and make this decision based primarily on sociocultural, religious, and/or familial norms.

Expectant parents' knowledge will be assessed via a Qualtrics survey. Participants will be recruited in the OB/GYN clinic sometime between their 24-28 week prenatal visit. We hope to accrue at least 680 participants for this study in order to achieve statistical significance and acquire a range of demographics. Expectant mothers and fathers (and single mothers) will be encouraged to participate.

This survey will assess their desire to get their child circumcised when they are born. Participants will be asked to list perceived risks and benefits of circumcision. This will hopefully allow us to see two things: if parents are aware and knowledgeable of the risks and benefits or circumcision, and what they perceive to be risky or beneficial from a medical standpoint.

Parents will be randomly given 1 of 2 pieces of information (1 per couple [or per single mother]; 1 control, 1 experiment) with different information about circumcision. We will see if there are any outcome differences based on which group the couple randomized into. Follow-up phone call will serve to assess outcome if baby was circumcised and any factors that led up to the decision. This will allow us to see if the AAP stance has any effect on decision making when we compare the control and experiment groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited from the Obstetrics clinic. All expectant parents of children are eligible to participate in this study. The study team will include those who do not know the sex of their baby and later exclude those who ultimately have girls from the final survey.

Exclusion Criteria:

* Exclusion is limited to parents with a child that has had a genital anomaly identified via ultrasound before the time of the research study, and parents that definitively know they are having girls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Number of children circumcised | 18 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States